CLINICAL TRIAL: NCT04664621
Title: HepQuant to Predict Hepatic Encephalopathy in Patients Who Receive Transjugular Intrahepatic Portosystemic Shunt (TIPS) for Refractory Ascites - a Pilot Study
Brief Title: HepQuant to Predict Hepatic Encephalopathy After TIPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant expired
Sponsor: Northwestern University (Other)
Collaborators: HepQuant, LLC (Industry)
Responsible Party: Principal Investigator, Justin Boike, Assistant Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00210205
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HepQuant Testing (Experimental)
  Interventions: Diagnostic Test: HepQuant

INTERVENTIONS:
Diagnostic Test: HepQuant — Patients undergoing TIPS procedure will receive a HepQuant test prior to and then after TIPS.

SUMMARY:
A pilot study to determine if a simple blood test can predict patients at risk for significant episodes of confusion and disorientation that can occur in patients who receive an artificial shunt through the liver to control complications of liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18 able to provide consent
* Subjects undergoing initial TIPS procedure for the primary indication of treatment of ascites

Exclusion Criteria:

* Prisoners
* Pregnant women
* Subjects undergoing TIPS placement as part of an investigational study outside of usual clinical care
* Subjects taking beta-blocker medications or angiotensin converting enzyme inhibitors
* Subjects with evidence of porto-systemic shunts present on imaging (eg splenorenal shunt)
* Subjects with calculated MELD score >12 based on most recent laboratory values before consent
* Subjects with prior history of overt hepatic encephalopathy (grade 3-4) that was primary reason for hospitalization. Episodes of hepatic encephalopathy that were the consequence of other precipitating event (such as variceal bleeding or infection) will not be considered exclusionary.
* Subjects with a known sensitivity to albumin preparations, any ingredient in the formulation, or components of the container
* Subjects unable to fast for >5 hours prior to the HepQuant administration or subjects who are unable to drink the oral dose of the cholate (~40mL of liquid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Onset of Hepatic Encephalopathy | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No